CLINICAL TRIAL: NCT01188876
Title: Phase I/II Study of Carboplatin and Pralatrexate in Patients With Recurrent Platinum-Sensitive Ovarian, Fallopian or Primary Peritoneal Cancer
Brief Title: Carboplatin/Pralatrexate in Recurrent Platinum-Sensitive Ovarian, Fallopian or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Marcela G. del Carmen, MD, MD, MPH, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-113
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: carboplatin; recurrent; platinum sensitive; pralatrexate
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Recurrence | interventions — Carboplatin; 10-propargyl-10-deazaaminopterin; Folic Acid; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin/Pralatrexate (Experimental)
  Interventions: Drug: carboplatin; Drug: pralatrexate; Drug: Folic Acid; Drug: Vitamin B12 Injection

INTERVENTIONS:
Drug: carboplatin — Given intravenously on Day 1 of each 28-day cycle
Drug: pralatrexate — Given intravenously on Day 1 and Day 15 of each 28-day cycle.
Drug: Folic Acid — Given orally on a daily basis starting 7 days before the first dose of pralatrexate and continuing until 30 days after the last dose of pralatrexate.
Drug: Vitamin B12 Injection — Given vitamin B12 injection no more than 10 weeks prior to the first dose of pralatrexate and every 8-10 weeks after the first dose of pralatrexate.

SUMMARY:
Pralatrexate is a type of antifolate drug which means is restrains the production of folic acid in the body. Folic acids are used by tumors to increase tumor cell growth and division. It is believed that reducing folic acid will hinder the rapid division of tumor cells, their growth and production. Carboplatin is an FDA approved chemotherapy drug for ovarian, fallopian tube and primary peritoneal cancer. Some antifolate drugs are used with other chemotherapy drugs to enhance cancer-fighting characteristics. It is believed that the study drug pralatrexate may improve the anti-tumor effect of carboplatin. In this research study we are looking for the highest dose of pralatrexate that can be given safely in combination with carboplatin.

DETAILED DESCRIPTION:
* Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects, not everyone who participates will receive the same dose of the study drug.
* Each study cycle will last 28 days. On Day 1, participants will receive carboplatin intravenously. On Days 1 and 15 of each cycle they will receive pralatrexate intravenously. Participants will also be asked to take folic acid orally on a daily basis starting 7 days before the first dose of pralatrexate and continuing until 30 days after the last dose of pralatrexate. They will also receive a vitamin B12 injection no more than 10 weeks prior to the first dose of pralatrexate and every 8-10 weeks after the first dose of pralatrexate.
* Participants will come to the clinic on Day 1 and 15 of each cycle and have the following tests/procedures performed: Medical history; Vital signs; Blood tests, assessment of the tumor (every two cycles) and an EKG (before the start of cycle 2).
* In addition, during Cycle 1, participants will come to the clinic weekly for blood tests.
* Pharmacokinetic (PK) blood samples (to monitor how the body absorbs and breaks down the study drug) will be done at the following time points during Cycle 1: Day 1-3 and Day 15-17.
* Participants will be asked to take the study drugs for up to 6 cycles. They may continue beyond 6 cycles as long as there is evidence that the tumor is not growing and they are not experiencing any unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with a platinum-sensitive recurrence of epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.
* The following histologic subtypes are eligible: papillary serous, endometrioid, mucinous, clear cell, adenocarcinomas, transitional, and mixtures of the above.
* Patients must have at least one measurable lesion according to RECIST criteria via CT or MRI scan. CT of the chest should be performed if any known disease is present in the chest. Pleural effusions, ascites, bone metastases, CA125 tumor markers, and lesions located in previously radiated areas are not considered measurable.
* Patients must have received a platinum-containing regimen at initial diagnosis.
* ECOG Performance Status of 0, 1 or 2
* Patients may have received up to 2 prior chemotherapy regimens in the recurrent cancer setting
* 18 years of age or older
* Life expectancy of greater than 12 weeks
* Baseline laboratory values must meet what is outlined in the protocol
* Patients must receive vitamin B12 and folic acid prior to starting treatment
* Complete recovery from previous chemotherapy or biologic therapy
* During the Phase II of the study, patients with significant ascites and/or pleural effusions will undergo consideration of drainage of these areas prior to starting carboplatin and pralatrexate.
* Women of childbearing potential must have a negative pregnancy test within 7 days prior to initiating chemotherapy on trial and must agree to practice effective method of birth control during the study and for six months after their last treatment.
* Patients must have a normal QTc interval

Exclusion Criteria:

* Prior pelvic radiotherapy to greater than 25% of bone marrow
* Any uncontrolled medical problem that in the opinion of the investigator would preclude safe administration of the study drugs.
* Past history of bone marrow transplantation or stem cell support
* Patient with known history of CNS metastasis is ineligible unless the patient has had treatment with surgery or radiation therapy, is neurologically stable, and does not require oral or intravenous corticosteroids or anticonvulsants.
* A history of prior malignancy except for adequately treated carcinoma in situ of the uterine cervix, incidental stage I endometrial cancer, basal cell or squamous cell skin cancer, or breast cancer (invasive or ductal carcinoma in situ) for which the patient has been disease-free for at least three years.
* Routine prophylactic use of G-CSF or GM-CSF within two weeks prior to study entry.
* Clinically significant cardiac disease
* Uncontrolled hypercalcemia or diabetes mellitus
* Any signs of intestinal obstruction that interfere with bowel function and/or nutrition
* Grade 2 or greater peripheral neuropathy
* Participation in an investigational study within three weeks prior to study entry.
* History of anaphylactic shock to prior platinum chemotherapy that would preclude safe administration of study carboplatin.
* History of psychiatric disability or other central nervous system disorder as judged by the principal investigator that would be considered significant and that would preclude informed consent, safe administration of study medications and affecting ability to comply with study procedures.
* Doses of ibuprofen in excess of 400mg QID.
* Interval cytoreductive surgery planned for while subject is on-study.
* Recurrence/progression within 6 months of receiving ay platinum regimen
* Patients with either pleural effusions or ascites are not eligible for Phase I of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcela G. del Carmen, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboplatin/Pralatrexate
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin/Pralatrexate
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 59 [39 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48
  Black or African American | 1
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) score
  * 0: Asymptomatic (Fully active, able to carry on all pre-disease activities without restriction)
  * 1: Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  Participants
    0 | 34
    1 | 16
Primary Site [Count of Participants; unit: Participants]
  Ovary | 34
  Fallopian Tube | 6
  Peritoneal | 5
  Other | 5
Histology Subtype [Count of Participants; unit: Participants]
  Serous | 30
  Endometrioid | 6
  Transitional Cell | 1
  Carcinosarcoma | 3
  Other | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose of Pralatrexate in combination with Carboplatin in this patient population. The unit is given in milligrams per square meter of body surface area. MTD was determined using a standard 3 + 3 dose escalation cohort, where 3 participants were enrolled on the starting dose of 30 mg/m2 and if no dose limiting toxicities (DLT) were experienced after a full cycle, 3 additional participants were enrolled at the next highest dose level. Each increase in dose level escalated the dose of Pralatrexate by 15 mg/m2. If during any dose level, 1 patient out of 3 develops a DLT, then 3 additional patients will be added to that dose level. If 2 out of the 3 patients placed on any dose level experience a DLT, the preceding dose is considered MTD. If 1/6 has a DLT, the next higher dose level will commence accrual (unless at level +5 and then accrual to the Phase I portion will stop). If ≥ 2 of 6 patients have a DLT, then the preceding dose will be considered MTD.
Time Frame: 1 year
Population: The participants that participated in the phase 1 dose escalation portion of the study
Measure: Number; unit: mg/m^2
Arm/Group | Carboplatin/Pralatrexate
Number analyzed (Participants) | 30
mg/m^2 | 105

2. Primary Outcome: Best Overall Response
Description: Summary of the best overall responses to treatment as assessed by RECIST (Response Evaluation Criteria In Solid Tumors).
  * Complete Response (CR): Disappearance of all target lesions
  * Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
  * Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Pralatrexate
Number analyzed (Participants) | 50
Participants
  Complete Response | 0
  Partial Response | 19
  Stable Disease | 24
  Progressive Disease | 5
  Unevaluable | 2

3. Secondary Outcome: Overall Survival
Description: The number of participants still alive at the given time points. The duration of time is measured from the start of treatment until death due to any cause, participants are censored at the date of the last evaluation. The number participants surviving at 6, 12, 18, and 24 months is shown.
Time Frame: 6, 12, 18, and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Pralatrexate
Number analyzed (Participants) | 50
Participants
  6 Months | 49
  12 Months | 49
  18 Months | 46
  24 Months | 33

4. Secondary Outcome: Progression Free Survival
Description: The number of participants alive and without disease progression at the given time-points. Time is measured from the start of treatment. Progression is defined as having at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Pralatrexate
Number analyzed (Participants) | 50
Participants
  3 Months | 44
  6 Months | 40

5. Secondary Outcome: Treatment Related Adverse Events
Description: Summary of the treatment related adverse events experienced by participants as assessed by Common Terminology Criteria for Adverse Events (CTCAE 4). Adverse events were assessed from the start of treatment until 30 days after the last dose of study drug.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Pralatrexate
Number analyzed (Participants) | 50
Participants
  Constipation | 2
  Mucositis | 13
  Nausea | 16
  Vomiting | 2
  Diarrhea | 1
  Anemia | 5
  Thrombocytopenia | 8
  Neutropenia | 6
  Febrile neutropenia | 2
  Hypersensitivity reaction | 17
  Hypomagnesemia | 3
  Pruritis | 1
  Rash | 3
  Fatigue | 15

6. Secondary Outcome: Maximum Concentration of Drug in Plasma (Cmax)
Description: The maximum concentration of Pralatrexate at day 1 and 15 among phase 1 participants dosed at 105 milligrams per square meter of body surface area (mg/m2). The concentration is given in micrograms per milliliter.
Time Frame: Day 1 and Day 15
Population: Participants that required a dose reduction due to an adverse event were excluded from the day 15 evaluation
Measure: Mean (95% Confidence Interval); unit: ug/ml
Arm/Group | Carboplatin/Pralatrexate
Number analyzed (Participants) | 17
ug/ml
  Day 1 | 23.87 [15.25 to 32.49]
  Day 15: number analyzed (Participants) | 9
  Day 15 | 17.61 [11.43 to 24.09]

7. Secondary Outcome: Area Under the Plasma Drug Concentration-Time Curve (AUC)
Description: Area under the plasma drug concentration-time curve (AUC) for phase 1 participants that were dosed at 105 mg/m2. AUC represents the actual body exposure to drug after administration of a dose of the drug and is expressed in micrograms * hour per milliliter (ug*h/mL).
Time Frame: Day 1 and Day 15
Population: Participants that required a dose reduction due to an adverse event were excluded from the day 15 evaluation
Measure: Mean (95% Confidence Interval); unit: ug*h/mL
Arm/Group | Carboplatin/Pralatrexate
Number analyzed (Participants) | 17
ug*h/mL
  Day 1 | 9.89 [7.20 to 12.58]
  Day 15 | 8.01 [6.19 to 9.83]

ADVERSE EVENTS:
Time Frame: Adverse events information was collected from the start of treatment until 30 days after the last dose of study medication was received (median duration of 7 months)
Arm/Group | Carboplatin/Pralatrexate
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 4/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Pralatrexate (N=50)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Thromboembolytic event (Blood and lymphatic system disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Pralatrexate (N=50)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 15 (19)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (3)
Allergic reaction (Immune system disorders) | 14 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Anaphylaxis (Immune system disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 16 (29)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bloating (Gastrointestinal disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Colonic obstruction (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 21 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (13)
Creatinine increased (Investigations) | 3 (4)
Depression (Psychiatric disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 11 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Fatigue (General disorders) | 40 (63)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (7)
Fever (General disorders) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (7)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (7)
Hypertension (Vascular disorders) | 5 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 22 (35)
Insomnia (Psychiatric disorders) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 24 (53)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 34 (61)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (4)
Neutrophil count decreased (Investigations) | 18 (25)
Pain (General disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Pelvic pain (Reproductive system and breast disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (12)
Platelet count decreased (Investigations) | 19 (36)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Upper respiratory infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 6 (10)
Vomiting (Gastrointestinal disorders) | 13 (19)
Watering eyes (Eye disorders) | 6 (6)
White blood cell decreased (Investigations) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes